CLINICAL TRIAL: NCT02889874
Title: A Randomised Phase III Trial of Adjuvant Radiation Therapy Versus Observation Following Breast Conserving Surgery and Endocrine Therapy in Patients With Molecularly Characterised Luminal A Early Breast Cancer
Brief Title: EXamining PErsonalised Radiation Therapy for Low-risk Early Breast Cancer
Acronym: EXPERT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Breast Cancer Trials, Australia and New Zealand (Other)
Collaborators: Breast International Group (Other); ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANZ1601/BIG 16-02; 2016-003527-33 (EudraCT Number)
Record Dates: First submitted 2016-08-25; First posted 2016-09-07 (Estimated); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Early Stage Breast Carcinoma
Keywords: Radiation therapy; omission; non-inferiority; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: Radiation Therapy & endocrine therapy (No Intervention): Patients randomized to Arm A will receive standard radiation therapy and adjuvant endocrine therapy (standard of care).
- B: No Radiation Therapy (ET only) (Experimental): Patients randomized to Arm B will not receive radiation therapy (omission of radiation therapy) and receive adjuvant endocrine therapy only.
  Interventions: Radiation: Omission of radiation therapy

INTERVENTIONS:
Radiation: Omission of radiation therapy — Omission of radiation therapy (adjuvant endocrine therapy only).
  Arms: B: No Radiation Therapy (ET only)

SUMMARY:
This is a randomised, phase III, non-inferiority trial evaluating radiation therapy versus observation following breast conserving surgery and planned endocrine therapy in patients with stage I breast cancer of luminal A subtype defined using the Prosigna (PAM50) Assay.

DETAILED DESCRIPTION:
Radiation therapy (RT) after breast conserving surgery to improve local control and survival is the current standard of care for patients with early breast cancer. However, breast cancer is a heterogeneous disease, and the absolute benefit of RT in individual patients varies substantially. Thus, a pressing priority in contemporary breast cancer management is to tailor RT utilisation to the individual recurrence risks by identifying patients who are unlikely to benefit from RT, thereby avoiding the morbidity and costs of over-treatment.

It is recognised that selected patients with early breast cancer are unlikely to derive benefits from RT after breast conserving surgery. However, randomised trials have not consistently identified patients who may safely omit RT using conventional clinical-pathologic characteristics.

Breast cancer intrinsic subtypes distinguished by gene expression profiling are shown to be associated with distinct clinical outcomes. There is substantial evidence supporting the clinical validity of multigene assays including the PAM50-based Prosigna Assay that identifies intrinsic subtypes and generates a Risk of Recurrence score (ROR) to quantify individual risks of distant relapse. Multigene assays are increasingly integrated into clinical practice to inform chemotherapy decision, highlighting their substantial practice changing potential in personalising the use of RT for early breast cancer.

A recent analysis of archived tumour specimens of 1,308 patients with early breast cancer has shown significant associations between local recurrence risk and the PAM50-defined intrinsic subtypes and ROR score. EXPERT presents a unique opportunity of clinical and public health importance to optimise personalised local therapy for early breast cancer through precise, individualised quantification of local recurrence risk to identify low-risk patients for whom RT after breast conserving surgery may be safely omitted.

ELIGIBILITY:
Inclusion Criteria: for registration in the study:

1. Female patients aged ≥ 50 years of any menopausal status.
2. Primary tumour characteristics as assessed by conventional histopathology:

   * Unifocal histologically confirmed invasive breast carcinoma
   * Maximum microscopic size ≤2 cm
   * Grade 1 or 2 histology
   * ER and PR positive in ≥10% of tumour cells in either the biopsy or breast conserving surgical specimen
   * HER2 negative on IHC (score 0 or 1+) or in situ hybridisation (ERBB2-amplification Ratio ERBB2/centromeres <2.0 or mean gene copy number <6). Equivocal IHC score (2+) must be assessed by ISH.
3. Primary tumour must be resected by breast conserving surgery with microscopically negative margins for invasive carcinoma and any associated ductal carcinoma in situ (no cancer cells adjacent to any inked edge/surface of specimen) or re-excision showing no residual disease.
4. Histologically confirmed negative nodal status determined by sentinel node biopsy or axillary dissection. Patients with pN0 (i+) disease are eligible for study participation (malignant cells ≤0.2 mm in regional lymph node(s) detected by hematoxylin-eosin (H&E) stain or IHC, including isolated tumour cells).
5. No evidence of distant metastasis.
6. Eligible for and willing to have adjuvant endocrine therapy.
7. ECOG performance status 0-2.
8. Availability of FFPE tumour block for Prosigna (PAM50) Assay.

For randomization to the study, patients must fulfill all of the following criteria:

1. Primary tumour characteristics as assessed by Prosigna (PAM50) Assay:

* Luminal A intrinsic subtype
* ROR score ≤60

Exclusion Criteria:

Any one of the following is regarded as a criterion for exclusion from the study:

1. Primary tumour characteristics:

   * Presence of multifocal or multicentric invasive carcinoma or ductal carcinoma in situ;
   * Evidence of clinical or pathologic T4 disease (extension to the chest wall, oedema or ulceration of skin, satellite skin nodules, inflammatory carcinoma);
   * The invasive component of the primary tumour is present as micro-invasion only;
   * Grade 3 histology;
   * Presence of lymphovascular invasion
2. Contra-indication or unwillingness to have adjuvant endocrine therapy.
3. Planned to receive adjuvant chemotherapy or biologic therapy after breast cancer surgery, i.e. any systemic therapy other than endocrine therapy is not permitted. Any therapy unrelated to cancer is permitted at the discretion of investigators.
4. Treated with neoadjuvant endocrine therapy, chemotherapy or biologic therapy prior to breast cancer surgery.
5. Prior breast or thoracic RT for any condition.
6. Pre-operative breast imaging evidence of disease aside from the primary carcinoma resected by breast conserving surgery.
7. Concurrent invasive breast carcinoma or ductal carcinoma in situ (synchronous or metachronous).
8. Prior diagnosis of invasive breast carcinoma or ductal carcinoma in situ in either breast irrespective of disease free interval.
9. A diagnosis of non-breast malignancy <5 years prior to randomisation with the following exceptions:

   * Patients who are diagnosed with carcinoma in situ of cervix, endometrium or colon; melanoma in situ; and basal or squamous cell carcinoma of the skin at any time prior to randomisation are not excluded from study participation.
   * Patients who are diagnosed with other non-breast malignancy ≥5 years prior to randomisation and without evidence of disease recurrence are not excluded from study participation.
10. Significant comorbidity precluding definitive RT for breast cancer (e.g. cardiovascular or pulmonary disease, scleroderma, systemic lupus erythematosus).
11. Life expectancy <10 years.
12. Documented mutation of BRCA1, BRCA2 or TP53, or at high genetic risk of breast cancer.
13. Pregnant or lactating patients.
14. Inability to be registered to the study ≤8 weeks after the last surgical procedure for breast cancer.
15. Inability to commence RT (if randomised to receive RT) no later than 12 weeks from the last surgical procedure for breast cancer.
16. Inability to provide written informed consent.
17. Psychiatric, addictive, or any disorder that precludes compliance with protocol requirements.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1167 (Estimated)
Dates: Start 2017-08-21 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Local recurrence rate after breast conserving surgery | 10 years
  The time from randomisation to the date of local recurrence (LR) as a site of first recurrence.

SECONDARY OUTCOMES:
Local-regional recurrence-free interval (LRRFI) | 10 years
  Time from randomisation to the date of local or regional recurrence as a site of first recurrence.
Distant recurrence-free interval (DRFI) | 10 years
  Time from randomisation to the date of distant recurrence, regardless of occurrence of any intervening local or regional recurrence, contralateral breast cancer or second (non-breast) primary invasive cancer.
Disease free survival including DCIS (DFS-DCIS) | 10 years
  Time from randomisation to date of first evidence of local (invasive breast carcinoma or DCIS), regional or distanct recurrence; contralateral breast cancer (invasive breast carcinoma or DCIS); second (non-breast) primary invasive cancer; or death.
Invasive disease free survival (iDFS) | 10 years
  Time from randomisation to date of first evidence of local (invasive breast carcinoma), regional or distanct recurrence; contralateral breast cancer (invasive breast carcinoma); second (non-breast) primary invasive cancer; or death.
Recurrence-free interval | 10 years
  Time from randomisation to the date of local, regional or distant recurrence as a site of first recurrence.
Overall survival (OS) | 10 years
  Time from randomisation to date of death from any cause.
Salvage RT or mastectomy rate | 10 years
  Time from randomisation to the receipt of salvage RT or mastectomy, individually and in combination (one or the other) as a composite endpoint.
Adverse events for patients | 5 years
  Adverse events during treatment (up to 5 years of endocrine therapy) assessed using NCI CTCAE v4.0.
Assessment of the impact of endocrine therapy | 5 years
  FACT-ES measure of endocrine symptoms.

OTHER OUTCOMES:
Quality of Life: Fear of recurrence | 5 years
  Fear of Cancer Recurrence Inventory
Quality of Life: Convenience of care | 5 years
  Visual Analogue Scales (convenience and impact of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Heath Badger, Study Director — Breast Cancer Trials, Australia and New Zealand; Boon H Chua, Prof, Study Chair — Prince of Wales Hospital
Locations (68):
- Argentina (3):
  - Sanatorio Britanico Rosariio, Rosario, Santa Fe Province
  - Instituto de Oncologia de Rosario, Santa Fe
  - Clinica Viedma, Sarmiento
- Australia (32):
  - The Canberra Hospital, Canberra, Australian Capital Territory
  - Macarthur Cancer Therapy Centre, Campbelltown, New South Wales
  - The Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St Vincent's Hospital, Sydney, Darlinghurst, New South Wales
  - Genesis Cancer Care Newcastle, Gateshead, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Mater Hospital Sydney, North Sydney, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Tamworth Rural Referral Hospital, Tamworth, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Genesis Cancer Care Wesley, Auchenflower, Queensland
  - Cancer Care Service - Bundaberg, Bundaberg, Queensland
  - Cancer Care Service - Hervey Bay, Bundaberg, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - GenesisCare Tennyson, Kurralta Park, South Australia
  - Ballarat Austin Radiation Oncology Centre, Ballarat, Victoria
  - Peter MacCallum Cancer Centre - Bendigo, Bendigo, Victoria
  - Peter MacCallum Cancer Centre - Moorabin, Bentleigh East, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Icon Cancer Centre Richmond, East Melbourne, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - GenesisCare Radiation Oncology Centre Frankston, Frankston, Victoria
  - University Hospital Geelong, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Ringwood Radiation Oncology Centre, Ringwood East, Victoria
  - Latrobe Regional Hospital, Traralgon, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Chile (5):
  - Hospital Luis Tisne Brousse, Santiago, Santiago Metropolitan
  - Centro Oncologico del Norte, Antofagasta
  - Hospital Sotero del Rio, Puente Alto
  - Hospital Barros Luco Trudeau, San Miguel
  - Instituto Nacional del Cancer, Santiago
- Ireland (2):
  - St Luke's Radiation Oncology Network, Dublin
  - University Hospital Galway, Galway
- Italy (2):
  - ASST Ospedale A. Manzoni UOS Oncologia, Lecco
  - Istituto Europeo di Oncologia, Milan
- New Zealand (4):
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
  - Palmerston North Hospital, Palmerston North
  - Wellington Hospital, Wellington
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Arnoa de Vilanova de Lleida, Lleida
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
- Switzerland (5):
  - Hirslanden Clinique des Grangettes, Chêne-Bougeries
  - Fondazione Oncologia Lago Maggiore, Locarno
  - Kantonsspital Winterthur, Winterthur
  - Brust-Zentrum AG Zurich, Zurich
  - Universitatsspital Zurich, Zurich
- Taiwan (10):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Chang-Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Anonymised Individual Patient Data (IPD) collected during the trial as per BCT Data Sharing Guidelines.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available for request after publication of the main/final study results; no end date.
Access Criteria: Subject to approval by Breast Cancer Trials: contact concept@bctrials.org.au for further information.
  Note that there may be additional circumstances preventing BCT from sharing requested data as outlined in the BCT Data Sharing Guidelines .

REFERENCES:
- See also: Breast Cancer Trials (formerly Australia & New Zealand Breast Cancer Trials Group — https://www.breastcancertrials.org.au/home